CLINICAL TRIAL: NCT01346540
Title: LUME-Lung 3: A Phase I/II Study of Continuous Oral Treatment With BIBF 1120 Added to Standard Gemcitabine/Cisplatin Therapy in First Line NSCLC Patients With Squamous Cell Histology
Brief Title: A Phase I/II Study of Continuous Oral Treatment With BIBF 1120 Added to Standard Gemcitabine/Cisplatin Therapy in First Line NSCLC Patients With Squamous Cell Histology.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1199.82; 2010-019707-32 (EudraCT Number: EudraCT)
Record Dates: First submitted 2011-04-19; First posted 2011-05-03 (Estimated); Results first posted 2018-09-10 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — nintedanib

ARMS (2):
- BIBF 1120 (Experimental): VEGF inhibitor
  Interventions: Drug: BIBF 1120
- Placebo (Placebo Comparator): BIBF 1120 placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BIBF 1120 — VEGF inhibitor
  Arms: BIBF 1120
Drug: Placebo — BIBF 1120 placebo
  Arms: Placebo

SUMMARY:
The LUME-Lung3 study is in 2 parts:

Run-in Phase I - Open label study to identify the Maximum Tolerated Dose of BIBF 1120 that can be added to standard first-line treatment with 3 weekly schedules of gemcitabine and cisplatin.

Phase II - Placebo controlled efficacy study of BIBF 1120 added to standard 3 weekly cycles of gemcitabine and cisplatin therapy in patients with at least Stable Disease after 2 previous courses of the chemotherapy

ELIGIBILITY:
Inclusion criteria:

Run-in Phase I

1. Histologically or cytologically confirmed diagnosis of stage IIIB/IV or recurrent Non Small Cell Lung Cancer (NSCLC) with squamous cell histology.
2. Measurable disease according to Response Evaluation Criteria in Solid Tumours ( RECIST 1.1).
3. Patient Eastern Cooperative Oncology Group (ECOG) score of 0-1.
4. Male or female patients age = 18 years.
5. Life expectancy of at least three (3) months.
6. Written informed consent in accordance with International Conference on Harmonisation - Good Clinical Practice (ICH-GCP) guidelines.

   Phase II - in addition to the above criteria:
7. Radiologically-confirmed at least stable disease after 2 prior cycles of cisplatin / gemcitabine chemotherapy.

Exclusion criteria:

1. Prior therapy for advanced or metastatic or recurrent Non Small Cell Lung Cancer (NSCLC). One prior adjuvant, neoadjuvant or adjuvant + neoadjuvant treatment is allowed if at least 12 months have elapsed between the end of the treatment and randomization
2. Prior treatment with other Vascular Endothelial Growth Factor Receptor (VEGFR) inhibitors (other than bevacizumab)
3. Any contraindications for treatment with gemcitabine and/or cisplatin.
4. Use of any investigational drug within 4 weeks of entering the 1199.82 study.
5. History of major thrombotic or clinically relevant bleeding event in the past 6 months.
6. Significant cardiovascular diseases (i.e. hypertension not controlled by medication.
7. Surgery within 4 weeks (except tumour biopsy) prior randomisation and incomplete wound healing.
8. Active brain metastases
9. Radiotherapy (except extremities) within 3 months prior to baseline imaging and radiotherapy for brain metastasis < 4 weeks prior baseline imaging.
10. Any other current malignancy or malignancy diagnosed within the past five (5) years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-04-14 (Actual); Primary Completion 2013-04-25 (Actual); Study Completion 2017-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (7):
- 1199.82.39004 Boehringer Ingelheim Investigational Site, Milan, Italy
- 1199.82.3102 Boehringer Ingelheim Investigational Site, Maastricht, Netherlands
- Spain (3):
  - 1199.82.3401 Boehringer Ingelheim Investigational Site, Barcelona
  - 1199.82.3406 Boehringer Ingelheim Investigational Site, Madrid
  - 1199.82.3410 Boehringer Ingelheim Investigational Site, Málaga
- United Kingdom (2):
  - 1199.82.4401 Boehringer Ingelheim Investigational Site, London
  - 1199.82.4402 Boehringer Ingelheim Investigational Site, Manchester

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Phase I was open-label, 3+3 dose-confirmation part of the trial aimed to confirm safety of nintedanib to a maximum dose of 200 milligram twice daily given in combination with the standard regimen of gemcitabine and cisplatin. Phase II was to be double-blind, randomised, placebo-controlled part, but this part of the trial was not conducted.
Groups:
- Nintedanib 150 Milligram: Patient received 150 milligram (mg) Nintedanib (BIBF 1120) soft gelatin capsules, administered orally twice daily until withdrawal criteria were fulfilled along with standard therapy of Gemcitabine and Cisplatin. Gemcitabine was administered as an intravenous infused dose of 1250 milligram per meter squared (mg/m2) on days 1 and 8 of each 21-day treatment cycle. Cisplatin was administered as an intravenous infused dose of 75 mg/m2 given on day 1 of each 21-day treatment cycle.
- Nintedanib 200 Milligram: Patient received 200 milligram (mg) Nintedanib (BIBF 1120) soft gelatin capsules, administered orally twice daily until withdrawal criteria were fulfilled along with standard therapy of Gemcitabine and Cisplatin. Gemcitabine was administered as an intravenous infused dose of 1250 milligram per meter squared (mg/m2) on days 1 and 8 of each 21-day treatment cycle. Cisplatin was administered as an intravenous infused dose of 75 mg/m2 given on day 1 of each 21-day treatment cycle.
Period: Overall Study
Arm/Group | Nintedanib 150 Milligram | Nintedanib 200 Milligram
Started | 4 | 12
Completed | 1 | 0
Not Completed | 3 | 12
Not completed — Progressive disease-RECIST 1.1 criteria | 3 | 8
Not completed — Adverse Event | 0 | 4

BASELINE CHARACTERISTICS:
Population: All patients who received at least one dose of any study medication were included in the Treated Set (TS)
Groups:
- Total: Total of all reporting groups
Arm/Group | Nintedanib 150 Milligram | Nintedanib 200 Milligram | Total
Number analyzed (Participants) | 4 | 12 | 16
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.5 (10.9) | 65.7 (5.0) | 65.4 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 4 | 11 | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs) During First Cycle for the Determination of the Maximum Tolerated Dose (MTD)
Description: The following drug-related adverse events (AEs) qualified as a DLT: Non-hematological toxicity - Common Terminology Criteria for Adverse Events (CTCAE) Grade ≥3 events excluding transient electrolyte abnormality, hyperuricemia and isolated elevation of gamma-glutamyl trans-peptidase. Gastrointestinal AEs (nausea, vomiting, diarrhoea, abdominal pain) or hypertension of CTCAE Grade ≥3 despite optimal supportive care/intervention. Alanine aminotransferase and or Aspartate aminotransferase elevation of CTCAE Grade ≥3. Haematological toxicity - Uncomplicated CTCAE Grade 4 neutropenia (that was not associated with fever of ≥38.5° Celsius) for >7 days (except during Cycle 1). CTCAE Grade 4 febrile neutropenia associated with fever ≥38.5º Celsius. A decrease in platelet levels to CTCAE Grade 4 or CTCAE Grade 3 associated with bleeding or requiring transfusion. The inability to resume nintedanib dosing within 14 days of stopping due to a drug-related AE was also considered a DLT.
Time Frame: Up to 21 days from first drug administration
Population: All patients who received at least one dose of nintedanib were included in the Safety Set.
Measure: Number; unit: Participants
Arm/Group | Nintedanib 150 Milligram | Nintedanib 200 Milligram
Number analyzed (Participants) | 4 | 12
Participants | 0 | 0

2. Secondary Outcome: Incidence of Adverse Events (AEs) According to the Common Terminology Criteria for Adverse Events (CTCAE) Version 3.00
Description: Incidence of adverse events (AEs) according to the Common Terminology Criteria for Adverse Events (CTCAE) Version 3.00 with grade 1-5.
Time Frame: From the first drug administration until 28 days after last study drug administration, up to 804 days
Population: Treated Set
Measure: Number; unit: Participants
Arm/Group | Nintedanib 150 Milligram | Nintedanib 200 Milligram
Number analyzed (Participants) | 4 | 12
Participants
  Grade 1 | 0 | 0
  Grade 2 | 0 | 0
  Grade 3 | 1 | 8
  Grade 4 | 3 | 2
  Grade 5 | 0 | 2

3. Primary Outcome: Maximum Tolerated Dose (MTD) of Nintedanib Added to Cisplatin/Gemcitabine Based on the Occurrence of DLTs During Treatment Cycle 1.
Description: The MTD was defined as the dose of nintedanib administered with gemcitabine/cisplatin at which no more than 1 of 6 patients experienced DLT (or one dose tier below that dose at which 2 or more of 6 patients experienced DLT) during the first 21-day treatment cycle. Any DLTs experienced after the start of the second treatment period were considered separately.
Time Frame: Up to 21 days from first drug administration
Population: All patients who received at least one dose of nintedanib were included in the Safety Set.
Measure: Number; unit: Milligram
Groups:
- Nintedanib 150/200 Milligram: Patient received 150 or 200 milligram (mg) Nintedanib (BIBF 1120) soft gelatin capsules, administered orally twice daily until withdrawal criteria were fulfilled along with standard therapy of Gemcitabine and Cisplatin. Gemcitabine was administered as an intravenous infused dose of 1250 milligram per meter squared (mg/m2) on days 1 and 8 of each 21-day treatment cycle. Cisplatin was administered as an intravenous infused dose of 75 mg/m2 given on day 1 of each 21-day treatment cycle.
Arm/Group | Nintedanib 150/200 Milligram
Number analyzed (Participants) | 16
Milligram | 200

ADVERSE EVENTS:
Time Frame: From the first drug administration until 28 days after last study drug administration, up to 804 days
Description: Adverse events ongoing from the end of the treatment visit were also captured.
Arm/Group | Nintedanib 150 Milligram | Nintedanib 200 Milligram
Serious Adverse Events (participants affected / at risk) | 2/4 | 5/12
Other Adverse Events (participants affected / at risk) | 4/4 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nintedanib 150 Milligram (N=4) | Nintedanib 200 Milligram (N=12)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Sudden death (General disorders) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 2
Respiratory tract infection (Infections and infestations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nintedanib 150 Milligram (N=4) | Nintedanib 200 Milligram (N=12)
Anaemia (Blood and lymphatic system disorders) | 2 | 3
Neutropenia (Blood and lymphatic system disorders) | 3 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 4
Atrial fibrillation (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Deafness (Ear and labyrinth disorders) | 1 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 3
Vertigo (Ear and labyrinth disorders) | 0 | 2
Blepharitis (Eye disorders) | 1 | 0
Lacrimation increased (Eye disorders) | 1 | 0
Visual acuity reduced (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Abdominal tenderness (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 8
Diarrhoea (Gastrointestinal disorders) | 4 | 5
Dyspepsia (Gastrointestinal disorders) | 2 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Gingival pain (Gastrointestinal disorders) | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 4 | 9
Retching (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 8
Asthenia (General disorders) | 1 | 6
Chest discomfort (General disorders) | 1 | 0
Chest pain (General disorders) | 1 | 2
Fatigue (General disorders) | 1 | 3
Malaise (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 1 | 1
Non-cardiac chest pain (General disorders) | 1 | 0
Oedema (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 1
Pyrexia (General disorders) | 0 | 3
Candida infection (Infections and infestations) | 0 | 1
Ear infection (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 1
Oral candidiasis (Infections and infestations) | 1 | 0
Oral herpes (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1
Rhinitis (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 2
Blood albumin decreased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 0 | 3
Blood lactate dehydrogenase increased (Investigations) | 0 | 1
Blood magnesium decreased (Investigations) | 0 | 1
Blood potassium decreased (Investigations) | 1 | 1
Blood sodium decreased (Investigations) | 0 | 1
Blood urea increased (Investigations) | 0 | 2
Blood uric acid increased (Investigations) | 0 | 2
Electrocardiogram QT prolonged (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 2
Haemoglobin decreased (Investigations) | 0 | 2
Monocyte count decreased (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 2
Platelet count decreased (Investigations) | 0 | 2
Weight decreased (Investigations) | 2 | 4
White blood cell count decreased (Investigations) | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 4 | 4
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2
Increased appetite (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 1
Dizziness postural (Nervous system disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 2 | 1
Lethargy (Nervous system disorders) | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 3
Anxiety (Psychiatric disorders) | 0 | 1
Depressed mood (Psychiatric disorders) | 1 | 0
Hallucination (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 4
Azotaemia (Renal and urinary disorders) | 0 | 1
Lower urinary tract symptoms (Renal and urinary disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 4
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1
Haemorrhage (Vascular disorders) | 1 | 0
Hot flush (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 4
Hypotension (Vascular disorders) | 0 | 1
Phlebitis (Vascular disorders) | 0 | 2
Thrombosis (Vascular disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
This trial was prematurely discontinued (Phase II was not conducted) following Sponsor's decision not to continue the trial in this indication.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.